CLINICAL TRIAL: NCT01110772
Title: Comparative Study of a Iodine + Cyanoacrylate (Integuseal) vs. Iodine and Isopropyl Alcohol in Skin Preparation for Prevention of Surgical Site Infections in Oncologic Surgery
Brief Title: Comparison of Iodine + Isopropyl Alcohol Versus Iodine + Antimicrobial Sealant for Skin Preparation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Kimberly-Clark de México (Unknown)
Responsible Party: Diana Vilar-Compte, MD, MsC, Departmentof Infectious Diseases. Instituto Nacional de Cancerología
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09003INI
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Surgical Site Infection
Keywords: Surgical site infection; Skin preparation; Cost analysis
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2-octyl cyanoacrylate (Experimental): As recommended, povidone iodine is used for skin antisepsis. After drying, a layer of cyanoacrylate is applied on the skin surface with the purpose of immobilizing skin bacteria.
  Interventions: Device: 2-octyl cyanoacrylate [InteguSEAL®]
- iodine povacrylex in isopropyl alcohol (Active Comparator): Iodine povacrylex in isopropyl alcohol (Duraprep 3M) This is considered a standard of care in our hospital as many other institutions. It's efficacy and safety have been demonstrated.
  Interventions: Device: Iodine povacrylex in isopropyl alcohol [Duraprep®, 3M]

INTERVENTIONS:
Device: 2-octyl cyanoacrylate [InteguSEAL®] — At operating room arrival prior to surgery, povidone-iodine is applied on the skin surface on concentric circles as recommended; after drying, the cyanoacrylate device is opened and a layer of the sealant is applied on the incision and skin site(IS100 for patients undergoing mastectomy, and IS200 for patients undergoing gynecologic or digestive tract surgeries).
  Other Names: InteguSEAL® (Kimberly Clark)
  Arms: 2-octyl cyanoacrylate
Device: Iodine povacrylex in isopropyl alcohol [Duraprep®, 3M] — At the operating room arrival a few minutes before the incision, cleansing and skin antisepsis is done with the prefilled device with iodine povacrylex in isopropyl alcohol as recommended by 3M.
  Other Names: Duraprep® (3M)
  Arms: iodine povacrylex in isopropyl alcohol

SUMMARY:
The purpose if this study is to determine whether a microbial sealant (iodine + cyanoacrylate) [InteguSEAL®, Kimberly-Clark] reduces surgical site infections when compared to iodine and isopropyl alcohol (povacrylex in isopropyl alcohol) [Duraprep®] in oncologic surgery.

DETAILED DESCRIPTION:
Patient's skin flora is a major source of pathogens, and microbial contamination of the surgical site is a likely precursor of SSI. A variety of skin products may be used, including iodophors, alcohol-containing products, and clorhexidine gluconate. Despite these perioperative tactics, bacteria continue to survive at the skin level and migrate to contaminate the wound.

A microbial sealant (InteguSEAL®, Kimberly-Clark) that uses cyanoacrylate to seal endogenous skin flora has demonstrated to reduce wound contamination. The efficacy of the microbial sealant in preventing SSI has been tested in cardiovascular surgery and open inguinal hernia repair, with a reduction on SSI rate when compared to standard skin preparations. This cyanoacrylate has not been tested in oncologic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years undergoing elective clean or clean-contaminated breast, gynecologic or digestive tract surgery
* Accepts to participate and signs the informed consent form
* Have a telephone number to be contacted after surgery

Exclusion Criteria:

* Previous allergy to one of the study products
* Two or more procedures in different anatomical sites at the same time / surgery (v.g. hysterectomy and mastectomy)
* Pregnancy
* Breast feeding
* Contaminated or infected surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | 30-45 days
  Patients we'll be followed prospectively by direct observation to evaluate if a surgical infection occurs. After 30 days of follow-up, patients will be classified as having or not a surgical site infection using the CDC criteria.

SECONDARY OUTCOMES:
Cost analysis | 30-45 days
  We'll be doing a cost-efectiveness analysis at the end of the study considering the treatment arm, complications developed from surgery to end of follow-up and costs for its treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Vilar-Compte, MD;MsC, Principal Investigator — Instituto Nacional de Cancerologia, Columbia
Locations (1):
- National Institute of Cancerology, Mexico City, Mexico City, Mexico